CLINICAL TRIAL: NCT00708123
Title: Comparison of the Clinical Efficacy From the Retention Phase of Fluoride Delivery of Fluoride Toothpastes Using an in Situ Caries Model
Brief Title: In Situ Caries of Fluoride Toothpastes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: T3157503
Record Dates: First submitted 2008-07-01; First posted 2008-07-02 (Estimated); Results first posted 2012-11-19 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-03

CONDITIONS: Healthy Subjects; Partial Denture Wearers; Caries
Keywords: remineralization; enamel; fluoride; caries; in situ
MeSH Terms: interventions — Fluorides

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Sodium Fluoride (NaF) toothpaste[1350 parts per million(ppm)F] (Active Comparator): Participants to brush their natural teeth twice daily with a full ribbon of NaF toothpaste (1350 ppm F as NaF) for one timed minute, after removing their partial denture from their mouth.
  Interventions: Drug: Sodium fluoride toothpaste
- NaF/Carbopol toothpaste (1400 ppm F) (Experimental): Participants to brush their natural teeth twice daily with a full ribbon of NaF and 0.5% carbopol toothpaste (1450 ppm F as NaF) for one timed minute, after removing their partial denture from their mouth.
  Interventions: Drug: Sodium fluoride toothpaste
- NaMFP/NaF toothpaste (1450 ppm F) (Active Comparator): Participants to brush their natural teeth twice daily with a full ribbon of NaMFPand NaF toothpaste (1450 ppm F - 1000 ppm F as NaMFP and 450 ppm F as NaF) for one timed minute, after removing their partial denture from their mouth.
  Interventions: Drug: Sodium fluoride toothpaste
- NaF toothpaste (250 ppm F) (Active Comparator): Participants to brush their natural teeth twice daily with a full ribbon of NaF toothpaste (250 ppm F as NaF) for one timed minute, after removing their partial denture from their mouth.
  Interventions: Drug: Sodium fluoride toothpaste
- Placebo toothpaste (0 ppm F) (Placebo Comparator): Participants to brush their natural teeth twice daily with a full ribbon of fluoride free toothpaste (0 ppm F) for one timed minute, after removing their partial denture from their mouth.
  Interventions: Drug: Placebo toothpaste

INTERVENTIONS:
Drug: Sodium fluoride toothpaste — Various fluoride toothpastes containing 1350 ppm F, 1450 ppm F, 1400 ppm F and 250 ppm F
  Other Names: Fluoride
  Arms: NaF toothpaste (250 ppm F); NaF/Carbopol toothpaste (1400 ppm F); NaMFP/NaF toothpaste (1450 ppm F); Sodium Fluoride (NaF) toothpaste[1350 parts per million(ppm)F]
Drug: Placebo toothpaste — Fluoride free toothpaste (0 ppm F)
  Arms: Placebo toothpaste (0 ppm F)

SUMMARY:
This study is to evaluate the effect of fluoride dentifrices on enamel with artificial caries lesions in an in situ model.

DETAILED DESCRIPTION:
Topical fluorides have been proven to be clinically effective in the prevention of dental caries. It is generally agreed that anti-caries effect of fluoride (F) is mainly by decreasing the rate of enamel demineralization and enhancing the rate of enamel remineralization. An in-situ Surface Micro-hardness (SMH) test is widely used to evaluate enamel demineralization and remineralization during the caries process. The aim of this study was to evaluate the efficacy of toothpaste formulations containing fluoride from different sources [sodium fluoride (NaF) and sodium monofluorophosphate (NaMFP)] using an in situ caries model.

ELIGIBILITY:
Inclusion Criteria

1. Consent: Demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form.
2. Age:Aged between 18 and 78 years.
3. Compliance:Understands and is willing, able and likely to comply with all study procedures and restrictions.
4. General Health:Good general health with (in the opinion of the investigator) no clinically significant and/or relevant abnormalities of medical history or oral examination that could interfere with subject safety during the study period.
5. Diagnosis: Oral - i. Currently living in the Indianapolis area which is a fluoridated community (1 ppm F). ii. Currently wearing a removable mandibular partial denture with sufficient room in the posterior buccal flange area to accommodate two enamel specimens (required dimensions 12 x 7 millimeters (mm). iii. Willing and capable of wearing their removable partial dentures 24 hours per day during each two week treatment period. iv.All restorations in a good state of repair.
6. Salivary Flow:Have a salivary flow rate in the range of normal values (unstimulated whole saliva flow rate = 0.2 ml/minute; gum base stimulated whole saliva flow rate = 0.8 ml/minute).

Exclusion Criteria

1. Pregnancy:Women who are known to be pregnant or who are intending to become pregnant over the duration of the study. No pregnancy test will be required.
2. Breast-feeding:Women who are breast-feeding.
3. Allergy/Intolerance: Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
4. Clinical Study/Experimental Medication:Participation in another clinical study or receipt of an investigational drug within 30 days of the first treatment visit, with the exception of study T3157495 where the wash in period prior to treatment is sufficient.
5. Antibiotics:Currently taking antibiotics or have taken antibiotics in the 2 weeks prior to the screening visit.
6. Fluoride:Taking fluoride supplements for medical reasons.
7. Dental Health: Current active caries or periodontal disease that may compromise the study or health of the subjects.
8. Personnel: a) A member of the site study staff, b) An employee of the sponsor, c) Any employee of any toothpaste manufacturer or their spouse or family member.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-11; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site.
Pre-assignment Details: Two days, prior to each treatment visit ,participants used a fluoride- free dentifrice twice daily to avoid any carry over effect.
Groups:
- Sodium Fluoride (NaF) Toothpaste[1350 Parts Per Million(Ppm)F]: Participants brushed their natural teeth twice daily with a full ribbon of NaF toothpaste (1350 ppm F as NaF) for one timed minute, after removing their partial denture from their mouth.
- NaF/Carbopol Toothpaste (1400 Ppm F): Participants brushed their natural teeth twice daily with a full ribbon of NaF and 0.5% carbopol toothpaste (1400 ppm F as NaF) for one timed minute, after removing their partial denture from their mouth.
- NaMFP/NaF Toothpaste (1450 Ppm F): Participants brushed their natural teeth twice daily with a full ribbon of NaMFP and NaF toothpaste (1450 ppm F - 1000 ppm F as NaMFP and 450 ppm F as NaF) for one timed minute, after removing their partial denture from their mouth.
- NaF Toothpaste (250 Ppm F): Participants brushed their natural teeth twice daily with a full ribbon of NaF toothpaste (250 ppm F as NaF) for one timed minute, after removing their partial denture from their mouth.
- Placebo Toothpaste (0 Ppm F): Participants brushed their natural teeth twice daily with a full ribbon of fluoride free toothpaste (0 ppm F) for one timed minute, after removing their partial denture from their mouth.
Period: Period 1
Arm/Group | Sodium Fluoride (NaF) Toothpaste[1350 Parts Per Million(Ppm)F] | NaF/Carbopol Toothpaste (1400 Ppm F) | NaMFP/NaF Toothpaste (1450 Ppm F) | NaF Toothpaste (250 Ppm F) | Placebo Toothpaste (0 Ppm F)
Started | 12 | 12 | 12 | 12 | 12
Completed | 12 | 11 | 11 | 11 | 12
Not Completed | 0 | 1 | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0
Period: Period 2
Arm/Group | Sodium Fluoride (NaF) Toothpaste[1350 Parts Per Million(Ppm)F] | NaF/Carbopol Toothpaste (1400 Ppm F) | NaMFP/NaF Toothpaste (1450 Ppm F) | NaF Toothpaste (250 Ppm F) | Placebo Toothpaste (0 Ppm F)
Started | 11 (Due to crossover design, different set of participants received this treatment compared to Period 1) | 12 (Due to crossover design,different set of participants received this treatment compared to Period 1) | 12 (Due to crossover design,different set of participants received this treatment compared to Period 1) | 11 (Due to crossover design, different set of participants received this treatment compared to Period 1) | 11 (Due to crossover design, different set of participants received this treatment compared to Period 1)
Completed | 10 | 12 | 12 | 10 | 11
Not Completed | 1 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0
Not completed — Other Reason | 1 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sodium Fluoride (NaF) Toothpaste[1350 Parts Per Million(Ppm)F] | NaF/Carbopol Toothpaste (1400 Ppm F) | NaMFP/NaF Toothpaste (1450 Ppm F) | NaF Toothpaste (250 Ppm F) | Placebo Toothpaste (0 Ppm F)
Started | 12 (Due to crossover design, different set of participants received this treatment compared to Period 2) | 10 (Due to crossover design, different set of participants received this treatment compared to Period 2) | 11 (Due to crossover design, different set of participants received this treatment compared to Period 2) | 12 (Due to crossover design, different set of participants received this treatment compared to Period 2) | 10 (Due to crossover design, different set of participants received this treatment compared to Period 2)
Completed | 12 | 10 | 10 | 11 | 10
Not Completed | 0 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0
Period: Period 4
Arm/Group | Sodium Fluoride (NaF) Toothpaste[1350 Parts Per Million(Ppm)F] | NaF/Carbopol Toothpaste (1400 Ppm F) | NaMFP/NaF Toothpaste (1450 Ppm F) | NaF Toothpaste (250 Ppm F) | Placebo Toothpaste (0 Ppm F)
Started | 10 (Due to crossover design, different set of participants received this treatment compared to Period 3) | 12 (Due to crossover design, different set of participants received this treatment compared to Period 3) | 10 (Due to crossover design, different set of participants received this treatment compared to Period 3) | 10 (Due to crossover design, different set of participants received this treatment compared to Period 3) | 11 (Due to crossover design, different set of participants received this treatment compared to Period 3)
Completed | 10 | 11 | 10 | 10 | 11
Not Completed | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0
Period: Period 5
Arm/Group | Sodium Fluoride (NaF) Toothpaste[1350 Parts Per Million(Ppm)F] | NaF/Carbopol Toothpaste (1400 Ppm F) | NaMFP/NaF Toothpaste (1450 Ppm F) | NaF Toothpaste (250 Ppm F) | Placebo Toothpaste (0 Ppm F)
Started | 10 (Due to crossover design, different set of participants received this treatment compared to Period 4) | 10 (Due to crossover design, different set of participants received this treatment compared to Period 4) | 11 (Due to crossover design, different set of participants received this treatment compared to Period 4) | 11 (Due to crossover design, different set of participants received this treatment compared to Period 4) | 10 (Due to crossover design, different set of participants received this treatment compared to Period 4)
Completed | 10 | 10 | 11 | 11 | 10
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: All randomized participants were included for baseline evaluation.
Arm/Group | All Study Participants
Number analyzed (Participants) | 60
Age Continuous [Mean (Standard Deviation); unit: years] | 67.31 (9.166)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 27
Region of Enrollment [Number; unit: participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Mean Percentage Surface Microhardness Recovery (%SMHR) of Enamel Specimens Exposed to NaF/Carbopol Toothpaste (1400 ppmF), NaF Toothpaste (1350ppmF) Compared to NaMFP/NaF Toothpaste (1450ppmF)
Description: %SMHR test was used to assess mineralization status of enamel specimens using a Wilson 2100 Hardness tester. %SMHR was determined by measuring the length of the indentations of enamel specimens. An increase in the indentation length compared to the baseline indicates softening while decrease in the indentation length represents rehardening of enamel surface. %SMHR was calculated from indentation values of enamel specimens at baseline (B), after intra-oral exposure (R) and after in-vitro demineralization (D) using formula: [(D-R)/ (D-B)]*100.
Time Frame: Baseline to 14 days
Population: Intent to treat population: All randomized participants who had at least one post baseline efficacy assessment. Missing data was not imputed. Due to subject drop outs, there are differences in the "n" per treatment group.
Measure: Least Squares Mean (Standard Error); unit: %SMHR
Groups:
- NaF Toothpaste (1350 Ppm F): Participants brushed their natural teeth twice daily with a full ribbon of NaF toothpaste (1350 ppm F as NaF) for one timed minute, after removing their partial denture from their mouth.
- NaMFP/NaF Toothpaste (1450 Ppm F): Participants brushed their natural teeth twice daily with a full ribbon of NaMFP and NaF toothpaste (1450 ppm F - 1000 ppm F as NaMFP and 450 ppm F as NaF) for one timed minute, after removing their partial dentures from their mouth.
Arm/Group | NaF/Carbopol Toothpaste (1400 Ppm F) | NaF Toothpaste (1350 Ppm F) | NaMFP/NaF Toothpaste (1450 Ppm F)
Number analyzed (Participants) | 54 | 53 | 54
%SMHR | 33.54 (1.72) | 35.23 (1.74) | 29.57 (1.72)
Statistical Analysis 1: Comparison: NaF/Carbopol Toothpaste (1400 Ppm F) vs NaMFP/NaF Toothpaste (1450 Ppm F); Null hypothesis was no difference between treatments being compared. Tests were 2-sided at 5% significance level; Test type: Superiority or Other; p = 0.0265, ANOVA — No adjustment was made for multiple comparisons as primary comparisons were pre-defined; The analysis included factors treatment, period and subject as a random effect; Adjusted mean difference = 3.97, 95% CI 2-sided [0.47 to 7.48] — Difference is first named treatment minus second named treatment such that a positive difference favors the first named treatment
Statistical Analysis 2: Comparison: NaF Toothpaste (1350 Ppm F) vs NaMFP/NaF Toothpaste (1450 Ppm F); Null hypothesis was no difference between treatments being compared. Tests were 2-sided at 5% significance level; Test type: Superiority or Other; p = 0.0017, ANOVA — No adjustment was made for multiple comparisons as primary comparisons were pre-defined; The analysis included factors as treatment, period and subject as a random effect; Adjusted mean difference = 5.66, 95% CI 2-sided [2.15 to 9.18] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Mean %SMHR of Enamel Specimens Exposed to NaF/Carbopol Toothpaste (1400 ppmF), NaF Toothpaste (1350ppmF), NaMFP/NaF Toothpaste (1450ppmF), NaF Toothpaste (250ppmF) and Placebo Toothpaste (0ppmF)
Description: as for outcome 1
Time Frame: Baseline to 14 days
Population: ITT population: All randomized participants who had at least one post baseline efficacy assessment. Missing data was not imputed. Due to drop outs, there were differences in the "n" per treatment group.
Measure: Least Squares Mean (Standard Error); unit: %SMHR
Groups:
- NaF/Carbopol Toothpaste (1400 Ppm F): Participants brushed their natural teeth twice daily with a full ribbon of NaF and 0.5% carbopol toothpaste (1450 ppm F as NaF) for one timed minute, after removing their partial denture from their mouth.
- NaF Toothpaste (1350ppm F): Participants brushed their natural teeth twice daily with a full ribbon of NaF toothpaste (1350 ppm F as NaF) for one timed minute, after removing their partial denture from their mouth.
Arm/Group | NaF/Carbopol Toothpaste (1400 Ppm F) | NaF Toothpaste (1350ppm F) | NaF Toothpaste (250 Ppm F) | NaMFP/NaF Toothpaste (1450 Ppm F) | Placebo Toothpaste (0 Ppm F)
Number analyzed (Participants) | 54 | 53 | 54 | 54 | 54
%SMHR | 33.54 (1.72) | 35.23 (1.74) | 24.98 (1.72) | 29.57 (1.72) | 22.05 (1.73)
Statistical Analysis 1: Comparison: NaF/Carbopol Toothpaste (1400 Ppm F) vs NaF Toothpaste (1350ppm F); Null hypothesis was no difference between treatments being compared. Tests were 2-sided at 5% significance level; Test type: Superiority or Other; p = 0.3413, ANOVA — No adjustment was made for multiple comparisons as the primary comparisons were pre-defined; ANOVA with factors for treatment, study period, and subject as random effect; Adjusted Mean DIfference = -1.69, 95% CI 2-sided [-5.19 to 1.80] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: NaF Toothpaste (1350ppm F) vs NaF Toothpaste (250 Ppm F); Null hypothesis was no difference between treatments being compared. Tests were 2-sided at 5% significance level; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustments made for multiple comparisons as the primary comparison was pre-specified; ANOVA with factors for treatment, study period, and subject as random effect; Adjusted Mean Difference = 10.26, 95% CI 2-sided [6.76 to 13.76] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: NaF Toothpaste (1350ppm F) vs Placebo Toothpaste (0 Ppm F); Null hypothesis was no difference between treatments being compared. Tests were 2-sided at 5% significance level; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment was made for multiple comparisons as the primary comparisons were pre-defined; ANOVA with factors for treatment, study period, and subject as random effect; Adjusted Mean Difference = 13.19, 95% CI 2-sided [9.69 to 16.68] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: NaF/Carbopol Toothpaste (1400 Ppm F) vs NaF Toothpaste (250 Ppm F); Null hypothesis was no difference between treatments being compared. Tests were 2-sided at 5% significance level; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment was made for multiple comparisons as the primary comparisons were pre-defined; ANOVA with factors for treatment, study period, and subject as random effect; Adjusted Mean Difference = 8.57, 95% CI 2-sided [5.09 to 12.05] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: NaF/Carbopol Toothpaste (1400 Ppm F) vs Placebo Toothpaste (0 Ppm F); Null hypothesis was no difference between treatments being compared. Tests were 2-sided at 5% significance level; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment was made for multiple comparisons as the primary comparisons were pre-defined; ANOVA with factors for treatment, study period, and subject (random effect); Adjusted Mean Difference = 11.50, 95% CI 2-sided [8.01 to 14.98] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: NaF Toothpaste (250 Ppm F) vs NaMFP/NaF Toothpaste (1450 Ppm F); Null hypothesis was no difference between treatments being compared. Tests were 2-sided at 5% significance level; Test type: Superiority or Other; p = 0.0104, ANOVA — No adjustment was made for multiple comparisons as the primary comparisons were pre-defined; ANOVA with factors for treatment, study period, and subject as random effect; Adjusted Mean Difference = -4.59, 95% CI 2-sided [-8.10 to -1.09] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: NaMFP/NaF Toothpaste (1450 Ppm F) vs Placebo Toothpaste (0 Ppm F); Null hypothesis was no difference between treatments being compared. Tests were 2-sided at 5% significance level; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment was made for multiple comparisons as the primary comparisons were pre-defined; ANOVA with factors for treatment, study period, and subject as random effect; Adjusted Mean Difference = 7.52, 95% CI 2-sided [4.04 to 11.01] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: NaF Toothpaste (250 Ppm F) vs Placebo Toothpaste (0 Ppm F); Null hypothesis was no difference between treatments being compared. Tests were 2-sided at 5% significance level; Test type: Superiority or Other; p = 0.0986, ANOVA — No adjustment was made for multiple comparisons as the primary comparisons were pre-defined; ANOVA with factors for treatment, study period, and subject as random effect; Adjusted Mean DIfference = 2.93, 95% CI 2-sided [-0.55 to 6.41] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Adjusted Mean Change From Baseline in Enamel Fluoride Uptake
Description: Enamel fluoride uptake was determined using the microdrill enamel biopsy technique. The amount of fluoride uptake by enamel was calculated based on the amount of fluoride (F) divided by the area of the enamel cores and expressed as ug F/cm2. The difference between treatments was calculated with respect to fluoride uptake by enamel.
Time Frame: Baseline to 14 days
Population: ITT population: All randomized participants who had a least one post baseline efficacy assessment. Missing data was not imputed. Due to drop outs, there were differences in the "n" per treatment group.
Measure: Least Squares Mean (Standard Error); unit: µg*F/cm^2
Groups:
- NaF/ Carbopol Toothpaste (1400 Ppm F): Participants brushed their natural teeth twice daily with a full ribbon of NaF and 0.5% carbopol toothpaste (1400 ppm F as NaF) for one timed minute, after removing their partial denture from their mouth.
Arm/Group | NaF/ Carbopol Toothpaste (1400 Ppm F) | NaF Toothpaste (1350ppm F) | NaF Toothpaste (250 Ppm F) | NaMFP/NaF Toothpaste (1450 Ppm F) | Placebo Toothpaste (0 Ppm F)
Number analyzed (Participants) | 54 | 53 | 54 | 54 | 54
µg*F/cm^2 | 1283.13 (71.53) | 1333.09 (72.08) | 680.20 (71.48) | 1086.39 (71.42) | 435.58 (71.54)
Statistical Analysis 1: Comparison: NaF/ Carbopol Toothpaste (1400 Ppm F) vs NaMFP/NaF Toothpaste (1450 Ppm F); Null hypothesis was no difference between treatments. Tests were 2-sided at 5% significance level; Test type: Superiority or Other; p = 0.0148, ANOVA — No adjustment was made for multiple comparisons as the primary comparisons were pre-defined; ANOVA with factors for treatment, study period, and subject as random effect; Adjusted Mean Difference = 196.74, 95% CI 2-sided [38.89 to 354.60] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: NaF Toothpaste (1350ppm F) vs NaMFP/NaF Toothpaste (1450 Ppm F); Null hypothesis was no difference between treatments being compared. Tests were 2-sided at 5% significance level; Test type: Superiority or Other; p = 0.0024, ANOVA — No adjustment was made for multiple comparisons as the primary comparisons were pre-defined; ANOVA with factors for treatment, study period, and subject as random effect; Adjusted Mean Difference = 246.70, 95% CI 2-sided [88.30 to 405.10] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: NaF/ Carbopol Toothpaste (1400 Ppm F) vs NaF Toothpaste (1350ppm F); Null hypothesis was no difference between treatments being compared. Tests were 2-sided at 5% significance level; Test type: Superiority or Other; p = 0.5328, ANOVA — No adjustment was made for multiple comparisons as the primary comparisons were pre-defined; ANOVA with factors for treatment, study period, and subject as random effect; Adjusted Mean Difference = -49.96, 95% CI 2-sided [-207.62 to 107.71] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: NaF Toothpaste (250 Ppm F) vs NaMFP/NaF Toothpaste (1450 Ppm F); Null hypothesis was no difference between treatments being compared. Tests were 2-sided at 5% significance level; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment was made for multiple comparisons as the primary comparisons were pre-defined; ANOVA with factors for treatment, study period, and subject as random effect; Mean Difference (Final Values) = -406.19, 95% CI 2-sided [-564.00 to -248.37] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: NaF/ Carbopol Toothpaste (1400 Ppm F) vs NaF Toothpaste (250 Ppm F); Null hypothesis was no difference between treatments being compared. Tests were 2-sided at 5% significance level; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment was made for multiple comparisons as the primary comparisons were pre-defined; ANOVA with factors for treatment, study period, and subject as random effect; Adjusted Mean Difference = 602.93, 95% CI 2-sided [445.97 to 759.90] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: NaF Toothpaste (1350ppm F) vs NaF Toothpaste (250 Ppm F); Null hypothesis was no difference between treatments being compared. Tests were 2-sided at 5% significance level; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment was made for multiple comparisons as the primary comparisons were pre-defined; ANOVA with factors for treatment, study period, and subject as random effect; Adjusted Mean Difference = 652.89, 95% CI 2-sided [495.05 to 810.72] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: NaF/ Carbopol Toothpaste (1400 Ppm F) vs Placebo Toothpaste (0 Ppm F); Null hypothesis was no difference between treatments being compared. Tests were 2-sided at 5% significance level; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment was made for multiple comparisons as the primary comparisons were pre-defined; ANOVA with factors for treatment, study period, and subject as random effect; Adjusted Mean Difference = 847.55, 95% CI 2-sided [690.54 to 1004.55] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: NaF Toothpaste (1350ppm F) vs Placebo Toothpaste (0 Ppm F); Null hypothesis was no difference between treatments being compared. Tests were 2-sided at 5% significance level; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment was made for multiple comparisons as the primary comparisons were pre-defined; ANOVA with factors treatment, period and subject as random effect; Adjusted Mean Difference = 897.50, 95% CI 2-sided [739.92 to 1055.08] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: NaMFP/NaF Toothpaste (1450 Ppm F) vs Placebo Toothpaste (0 Ppm F); Null hypothesis was no difference between treatments being compared. Tests were 2-sided at 5% significance level; Test type: Superiority or Other; p < 0.0001, ANOVA — No adjustment was made for multiple comparisons as the primary comparisons were pre-defined; ANOVA with factors for treatment, study period, and subject as random effect; Adjusted Mean Difference = 650.80, 95% CI 2-sided [493.61 to 808.00] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: NaF Toothpaste (250 Ppm F) vs Placebo Toothpaste (0 Ppm F); Null hypothesis was no difference between treatments being compared. Tests were 2-sided at 5% significance level; Test type: Superiority or Other; p = 0.0024, ANOVA — No adjustment was made for multiple comparisons as the primary comparisons were pre-defined; ANOVA with factors for treatment, study period, and subject as random effect; Adjusted Mean Difference = 244.62, 95% CI 2-sided [87.62 to 401.61] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: All AEs encountered or spontaneously reported following administration of any investigational product (including washout product), or for up to 5 days after the last administration of investigational product were recorded.
Arm/Group | NaF/ Carbopol Toothpaste (1400 Ppm F) | NaF Toothpaste (1350ppm F) | NaMFP/NaF Toothpaste (1450 Ppm F) | NaF Toothpaste (250 Ppm F) | Placebo Toothpaste (0 Ppm F)
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/54 | 0/55 | 0/56 | 0/54
Other Adverse Events (participants affected / at risk) | 4/56 | 4/54 | 1/55 | 1/56 | 2/54
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NaF/ Carbopol Toothpaste (1400 Ppm F) (N=56) | NaF Toothpaste (1350ppm F) (N=54) | NaMFP/NaF Toothpaste (1450 Ppm F) (N=55) | NaF Toothpaste (250 Ppm F) (N=56) | Placebo Toothpaste (0 Ppm F) (N=54)
Nasopharyngitis (Infections and infestations) | 4 (4) | 4 (4) | 1 (1) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.